CLINICAL TRIAL: NCT00200707
Title: Intracoronary Injection of Autologous Bone Marrow Mononuclear Cells for Severe Myocardial Infarction
Brief Title: BONAMI (BOne Marrow in Acute Myocardial Infarction)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/03/2-B
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Acute and Severe Myocardial Infarction
Keywords: Cell therapy; bone marrow mononuclear cells; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The treatment group (Experimental): Intracoronary Injection of Autologous Bone Marrow Mononuclear C
  Interventions: Procedure: Intracoronary injection of autologous bone marrow mononuclear cells
- the control group (No Intervention)

INTERVENTIONS:
Procedure: Intracoronary injection of autologous bone marrow mononuclear cells
  Arms: The treatment group

SUMMARY:
Emerging evidence suggests that stem cells and progenitor cells derived from bone marrow can be used to improve cardiac function in patients after acute myocardial infarction. In this randomised trial, we aim to assess whether intracoronary transfer of autologous bone-marrow cells could improve myocardial viability at 3 and 12 months' follow-up.

DETAILED DESCRIPTION:
After successful percutaneous coronary intervention (PCI) for acute myocardial infarction, 100 patients are randomly assigned to either a control group (n=50) who receives an optimal medical treatment, or a bone-marrow-cell group (n=50) who receives an optimal medical treatment and intracoronary transfer of autologous bone-marrow cells 7•10 days after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18-75 years.
* Acute myocardial infarction
* Absence of viability in the infarcted zone and LVEF <45%.

Exclusion Criteria:

* History of prior myocardial infarction
* Significant stenosis in another coronary territory than the acutely treated vessel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2004-12; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in Myocardial viability evaluated by thallium scintigraphy (3 months and 1 year) | after 3 months and 1 year of treatment

SECONDARY OUTCOMES:
Left ventricle ejection fraction (LVEF) evaluated by radionuclide ventriculography, (3 and 12 months) and by echography (1, 3, 6, and 12 months). Segmental EF and myocardial viability evaluated by MRI (3 months) | after 1,3,6 ,12 months of treatment
Correlation with biological parameters (hematopoietic stem cell number, etc.) at the time of cell injection

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LEMARCHAND, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Manrique A, Lemarchand P, Delasalle B, Lairez O, Sportouch-Duckan C, Lamirault G, Le Corvoisier P, Neuder Y, Richardson M, Lebon A, Roncalli J, Piot C, Trochu JN, Teiger E, Hossein-Foucher C, Le Tourneau T. Predictors of ventricular remodelling in patients with reperfused acute myocardial infarction and left ventricular dysfunction candidates for bone marrow cell therapy: insights from the BONAMI trial. Eur J Nucl Med Mol Imaging. 2016 Apr;43(4):740-8. doi: 10.1007/s00259-015-3279-z. Epub 2015 Dec 15. PMID 26666236
- [Derived] Roncalli J, Mouquet F, Piot C, Trochu JN, Le Corvoisier P, Neuder Y, Le Tourneau T, Agostini D, Gaxotte V, Sportouch C, Galinier M, Crochet D, Teiger E, Richard MJ, Polge AS, Beregi JP, Manrique A, Carrie D, Susen S, Klein B, Parini A, Lamirault G, Croisille P, Rouard H, Bourin P, Nguyen JM, Delasalle B, Vanzetto G, Van Belle E, Lemarchand P. Intracoronary autologous mononucleated bone marrow cell infusion for acute myocardial infarction: results of the randomized multicenter BONAMI trial. Eur Heart J. 2011 Jul;32(14):1748-57. doi: 10.1093/eurheartj/ehq455. Epub 2010 Dec 2. PMID 21127322